CLINICAL TRIAL: NCT00386685
Title: Open Label, Uncontrolled Study of XRP9881 in Combination With Trastuzumab (Herceptin®) in Patients With HER2 Positive Metastatic Breast Cancer (MBC)
Brief Title: XRP9881 in Combination With Trastuzumab in Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Trial Transparency Team, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCD6595; XRP9881
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2011-04-12 (Estimated); Status verified 2011-04

CONDITIONS: Breast Neoplasms
Keywords: Cancer; Breast; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — larotaxel; Trastuzumab

INTERVENTIONS:
Drug: larotaxel (XRP9881) — intravenous administration
Drug: trastuzumab — intravenous administration

SUMMARY:
The primary objective of the study is to assess the activity of XRP9881 in combination with trastuzumab.

The secondary objectives are safety and pharmacokinetic interaction

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer (MBC)
* HER2 (Human Epidermal Growth Factor Receptor 2) positive: FISH (Fluorescent In Situ Hybridization) positive or IHC (Immunohistochemistry) 3+
* Measurable disease according to Response Evaluation Criteria In Solid Tumors (RECIST)
* Adequate organs functions

Exclusion Criteria:

* More than one previous chemotherapy regimen for metastatic disease
* Cardiac dysfunction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Response rate (best overall response under treatment) | study period

SECONDARY OUTCOMES:
Incidence of grade 3-4 toxicities, pharmacokinetic interaction | study period

CONTACTS AND LOCATIONS:
Overall Officials: Henri Roche, PhD, Principal Investigator — Institut Claudius Regaud - Toulouse - France
Locations (4):
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland